CLINICAL TRIAL: NCT05800119
Title: Exemption: Perception of Mental Disorders
Brief Title: An Intervention to Correct Dualistic Reasoning About the Effectiveness of Psychotherapy for Biologically Caused Mental Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2000025071; 2000029423 (Other: Yale University Institutional Review Board)
Record Dates: First submitted 2023-03-22; First posted 2023-04-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were not made aware of the condition they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Brain-level condition (Experimental): Participants assigned to this condition received a brief reading passage (126 words) that provided psychoeducation about how psychotherapy can change the brain of those with depression, and specifically how psychotherapy can change the functioning of the prefrontal cortex and the amygdala, and affect neurotransmitters.
  Interventions: Behavioral: Brain-level condition
- Mind-level condition (Active Comparator): Participants assigned to this condition received a brief reading passage (115 words) that provided psychoeducation about the effectiveness of psychotherapy for depression, and specifically how psychotherapy can improve maladaptive thought processes and teach people with depression how to regulate negative emotions.
  Interventions: Other: Mind-level condition
- Control condition (No Intervention): Participants assigned to this condition received no additional materials.

INTERVENTIONS:
Behavioral: Brain-level condition — Participants will receive a brief reading passage about the neurobiological effects of psychotherapy.
  Arms: Brain-level condition
Other: Mind-level condition — Participants will receive an active control consisting of a brief reading passage about the effectiveness of psychotherapy.
  Arms: Mind-level condition

SUMMARY:
The goal of this clinical trial is to test in three samples, including sample 1: lay people without reported depression symptoms, sample 2: lay people with reported depression symptoms and sample 3: mental health clinicians. The main questions it aims to answer are: 1) do each of these populations show a bias against psychotherapy wherein they judge psychotherapy to be less effective, relative to baseline ratings, when a mental illness (i.e., depression) is attributed to biological factors, 2) whether an intervention emphasizing the neurobiological effects of psychotherapy can remove this bias against psychotherapy for biologically-caused mental disorders, and 3) whether this intervention is more effective compared to an active control intervention that emphasizes the effectiveness of psychotherapy, but not its neurobiological effects. Participants will

* rate the effectiveness of psychotherapy for depression before and after learning about the biological causes of depression
* be assigned to one of three conditions: 1) an intervention condition where participants will receive a brief reading passage (approximately 126 words in length) providing psychoeducation about how psychotherapy changes the brain of an individual with depression, or 2) an active control condition where participants will receive a reading passage (approximately 115 words) emphasizing the effectiveness of psychotherapy, or 3) a control condition where they will receive no additional materials
* as a secondary outcome, participants will also rate the effectiveness of medication for depression, before and after learning about the biological causes of depression

DETAILED DESCRIPTION:
Overview: Previous studies showed that biological explanations for mental disorders, which are popularizing, cause laypeople and clinicians to judge that psychotherapy is less effective. This could be clinically detrimental, as the combination of pharmacotherapy and psychotherapy is often optimal. Objective: This study tests a "de-biasing" intervention developed to counteract the flawed dualistic belief that activities perceived as occurring in the mind (e.g., psychotherapy) do not necessarily affect the brain. Design, Setting, Participants: This survey was conducted between September 10, 2020 and April 2, 2022 through Qualtrics.com over laypeople with and without symptoms of depression, and licensed clinicians in the U.S. Participants were randomly assigned to either an intervention condition explaining how psychotherapy results in brain-level changes, an active control condition explaining the effectiveness of psychotherapy but not its biological mechanisms, or a control condition with no intervention. Main Outcome Measures: Participants rated the efficacy of psychotherapy for biologically caused depression before and after being assigned to one of the three conditions. It was hypothesized that the dualism intervention would increase ratings of the effectiveness of psychotherapy, even after participants learned about the biological causes of depression. It was also expected that this intervention would increase psychotherapy ratings more than the active control materials that also emphasized the effectiveness of psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participation was open to individuals in the US
* For sample 1, lay people without reported depression symptoms, there was no specific inclusion criteria
* For sample 2, lay people with reported depression symptoms, participants were included if they indicated via Amazon Mechanical Turk Toolkit that they experienced symptoms of depression
* For sample 3, mental health clinicians, participants were included if they indicated that they were a practicing mental health clinician in the United States

Exclusion Criteria:

* For lay people without reported depression symptoms, the only exclusion criteria was age (i.e., no participants under 18 years of age)
* For lay people with reported depression symptoms, participants were excluded if they scored < 14 on the Beck Depression Inventory-II (BDI-II), indicating no depression symptoms
* For mental health clinicians, participants were excluded if they indicated that they were not currently licensed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1243 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-04-02 (Actual)

PRIMARY OUTCOMES:
Change in beliefs about the effectiveness of psychotherapy from baseline to after learning about the biological causes of depression, as measured by two survey questions taken at pretest and at post-test | Pretest and post-test, both measures completed during an approximately 10-minute survey
  This outcome is measured with two questions, both on a 1-7 rating scale. The questions measure participants' beliefs about the effectiveness of psychotherapy. These two questions were asked on an online survey where participants completed the questions at pretest (before participants learned about the biological causes of depression, and were assigned to one of the three conditions) and at post-test. The questions were as follows: 1) "how effective would psychotherapy treatment be at addressing what might be the causes of depression? From 1 "not at all effective" to 7 "extremely effective" and 2) "how likely is it that symptoms will improve with psychotherapy treatment? From 1 "no improvement" to 7 "full recovery with no remaining symptoms." These questions were averaged to create a composite pretest and post-test psychotherapy effectiveness score. The change in mean scores from pretest to post-test will be the outcome of interest.

SECONDARY OUTCOMES:
Change in beliefs about the effectiveness of medication from baseline to after learning about the biological causes of depression, as measured by two survey questions taken at pretest and at post-test | Pretest and post-test, both measures completed during an approximately 10-minute survey
  This outcome is measured with two questions, both on a 1-7 rating scale. The questions measure participants' beliefs about the effectiveness of medication. These two questions were asked on an online survey where participants completed the questions at pretest (before participants learned about the biological causes of depression, and were assigned to one of the three conditions) and at post-test. The questions were as follows: 1) "how effective would medication treatment be at addressing what might be the causes of depression? From 1 "not at all effective" to 7 "extremely effective" and 2) "how likely is it that symptoms will improve with medication treatment? From 1 "no improvement" to 7 "full recovery with no remaining symptoms." These questions were averaged to create a composite pretest and post-test medication effectiveness score. The change in mean scores from pretest to post-test will be the secondary outcome of interest.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No